CLINICAL TRIAL: NCT04461626
Title: Prospective Multi-centre Outcomes Study of Persona Knee System in Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSA2014-02K
Record Dates: First submitted 2020-07-01; First posted 2020-07-08 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persona fixed bearing knee system: Persona fixed bearing knee system (All patients will received Persona fixed bearing knee system)
  Interventions: Device: Persona fixed bearing knee system (All patients will receive Persona fixed bearing knee system)

INTERVENTIONS:
Device: Persona fixed bearing knee system (All patients will receive Persona fixed bearing knee system)

SUMMARY:
This is a prospective, multi-centre, non comparative, post market clinical follow-up study involving orthopaedic surgeons skilled in TKA and experienced implanting the devices included in this study.

DETAILED DESCRIPTION:
The objectives of the study are to document the implant survivorship and clinical outcomes data for the Persona fixed bearing implants used in primary total knee arthroplasty (TKA). The study will include a maximum of 20 centres and up to 1000 implanted knees. Each centre may enrol up to a maximum of 100 implanted knees to permit assessment of the consistency of outcomes across a variety of investigators and clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years old, inclusive
* Qualifies for a primary TKA based on physical exam and medical history, including diagnosis of severe knee pain and disability due to at least one of the following:

  1. Rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis.
  2. Collagen disorders and/ or avascular necrosis of femoral condyle.
  3. Post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy.
  4. Moderate valgus, varus or flexion deformities.
  5. The salvage of previously failed surgical attempts that did not include partial or total knee arthroplasty of the ipsilateral knee.
* Participated in a study-related informed consent process.
* Willing and able to provide written informed consent by signing and dating the IRB/EC approved informed consent form.
* Willing and able to complete scheduled study procedures and follow-up evaluations.
* Independent of study participation, patient is a candidate for commercially available Persona fixed bearing knee system implanted in accordance with product labelling.

Exclusion Criteria:

* Currently participating in any other surgical intervention studies or pain management studies.
* Previous history of infection in the affected joint and/or other local/systemic infection that may affect the prosthetic joint.
* Insufficient bone stock on femoral or tibial surfaces/
* Skeletal immaturity
* Neuropathic arthropathy
* Any loss of musculature or neuromuscular disease that compromises the affected limb.
* Stable, painless arthrodesis in a satisfactory functional position.
* Severe instability secondary to the absence of collateral ligament integrity.
* Rheumatoid arthritis accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin.
* Known or suspected sensitivity or allergy to one or more of the implant materials.
* Pregnant or considered a member of a protected population (e.g. prisoner, mentally incompetent, etc.)
* Previously received partial or total knee arthroplasty for the ipsilateral knee.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients who require primary TKA and satisfy eligible criteria outlined in this section. In order to avoid potential selection bias, each investigator will offer study participation to each consecutive eligible patient presenting as a candidate for primary TKA using the Persona fixed bearing knee system.
Sampling Method: Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Implant Survivorship | Up to 5 years post surgery
  Implant survivorship based on removal of the study device and will be summarized using Kaplan-Meier analysis
Adverse Events (Safety) | Up to 5 years post surgery
  Safety based on incidence and frequency of adverse events
Clinical Performance | Up to 5 years post surgery
  Clinical Performance measured by overall pain and function and qualify of life Measured using EQ5D questionnaire and Knee Society Score
Clinical Performance | Up to 5 years post surgery
  Clinical Performance measured by physician assessment of radiographs form. Data collected include the position and assessment of the radiographs of the operated knee

CONTACTS AND LOCATIONS:
Overall Officials: Myung Chul Lee, Principal Investigator — Seoul National University Hospital
Locations (18):
- Fremantle Hospital, West Perth, Australia
- India (5):
  - Fortis Health Care, Bangalore, Bangalore
  - Sant Parmanand Hospital, Delhi
  - All India Institute of Medical Sciences, Delhi
  - Landmark Hospitals, Hyderabad
  - Deenanath Mangeshkar Hospital, Pune
- Japan (2):
  - Kochi University Hospital, Kochi
  - Nihon University Hospital, Tokyo
- Waikato Hospital, Hamilton, Waikato Region, New Zealand
- Singapore General Hospital, Singapore, Singapore
- South Korea (8):
  - GangNeung Asan Hospital, Gangneung
  - Chonnam National University Hwasun Hospital, Hwasun
  - Chungang University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Asan Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No